CLINICAL TRIAL: NCT03653494
Title: Department of Anesthesiology in Shenzhen People's Hospital
Brief Title: the Clinicaltrail of the Effection Which of Phrenic Block Using in Non-intubated Video-assisted Thoracoscopic Surgery
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: daizhongliang-02
Record Dates: First submitted 2018-07-16; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-05

CONDITIONS: Phrenic Nerve Paralysis
Keywords: non-intubated general anaesthesia; video-assisted thoracoscopic surgery; phrenic block

STUDY DESIGN:
Intervention Model Description: 1. Put 80 patients divided into group S（non-intubated general anesthesia combine with Paravertebral blocks、surface spray anesthesia and Vagus block） and group D（non-intubated general anesthesia combine with Paravertebral blocks、surface spray anesthesia、Vagus block and Phrenic block）randomly.
  2. Compare the volume of anesthetic drugs between the two groups.
  3. If the date of group S greater than group D，it shows that the effect of anesthetic effect of group D is better than group S.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Volunteers and data collectors was masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- phrenic block group (Experimental): non-intubated general anesthesia combine with Paravertebral blocks、surface spray anesthesia、Vagus block and Phrenic block
  Interventions: Procedure: phrenic block
- Control group (Active Comparator): non-intubated general anesthesia combine with Paravertebral blocks、surface spray anesthesia and Vagus block
  Interventions: Procedure: no phrenic block

INTERVENTIONS:
Procedure: phrenic block — phrenic block by 1% ropivacaine 5ml
  Arms: phrenic block group
Procedure: no phrenic block — no phrenic block
  Arms: Control group

SUMMARY:
Putting 80 patients divided into group S（non-intubated general anesthesia combine with Paravertebral blocks、surface spray anesthesia and Vagus block） and group D（non-intubated general anesthesia combine with Paravertebral blocks、surface spray anesthesia、Vagus block and Phrenic block）randomly,compare the volume of anesthetic and the number of increasing anesthetic during operation were compared between the two groups.If the date of group S greater than group D，it shows that the effect of anesthetic effect of group D is better than group S.

DETAILED DESCRIPTION:
1. Put 80 patients divided into group S（non-intubated general anesthesia combine with Paravertebral blocks、surface spray anesthesia and Vagus block） and group D（non-intubated general anesthesia combine with Paravertebral blocks、surface spray anesthesia、Vagus block and Phrenic block）randomly.
2. Compare the volume of anesthetic drugs between the two groups.
3. If the date of group S greater than group D，it shows that the effect of anesthetic effect of group D is better than group S.

ELIGIBILITY:
Inclusion Criteria:

* The patient agreed to perform non-intubated video-assisted thoracoscopic surgery, and informed the possibility of intraoperative tracheal intubation or thoracotomy.
* No conventional anesthesia contraindication, no history of thoracic surgery, good cardiopulmonary function.
* There is no severe adhesion and calcification in the thoracic cavity, and no artificial pneumothorax is affected.
* the patient has no serious anxiety or depression.
* Small surgical trauma, simple steps, short time.

Exclusion Criteria:

* Mallampati≥3.
* BMI≥26 kg/m2.
* Hemodynamic instability.
* INR≥1.5.
* Respiratory infection, persistent cough or airway mucus hypersecretion, high risk of reflux.
* nervous system disease,such as seizure or brain edema.
* Extensive pleural adhesions or once chest surgery.
* PaO2<60mmHg or PaCO2>50 mmHg.
* Central hypopnea syndrome.
* Lung isolation should be used to protect the healthy side of the lung.
* Complicated operation, large trauma, long time, lack of experience or poor cooperation in the surgical team.
* Contraindications to local anesthetic.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
the volume of anesthetic drugs | the time of operation， an average of 4 hours
  the volume of anesthetic drugs including sevoflurane,propofol and opioids during the operation

SECONDARY OUTCOMES:
the time to get out of bed after surgery | two days after surgery
  note the time to get out of bed after surgery
the cost of hospitalization | the time of hospitalization， an average of 7 days
  note the the cost of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Dai Z Liang, Doctor, Study Chair — Shenzhen People's Hospital
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No